CLINICAL TRIAL: NCT06695312
Title: Effect of High Tone Power Therapy on Neck Pain and Proprioception in Cervical Radiculopathy Patients
Brief Title: High Tone Power Therapy on Neck Pain and Proprioception in Cervical Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Assistant Professor of Neurology and Neurosurgery Faculty of Physical Therapy October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/0053400
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Other): the study group received the selected exercise program in addition to High Tone Power Therapy
  Interventions: Other: selected exercise program; Device: High Tone Power Therapy
- control group (Other): therapeutic ultrasound, Static neck exercise,
  Interventions: Other: selected exercise program

INTERVENTIONS:
Other: selected exercise program — therapeutic ultrasound, Static neck exercise
Device: High Tone Power Therapy — High Tone Power Therapy delivered in cervical region 3 times per week for four weeks
  Arms: study group

SUMMARY:
To investigate the Effect of High Tone Power Therapy on Neck Pain and Proprioception in Cervical Radiculopathy Patients.

DETAILED DESCRIPTION:
Forty two patients with Cervical Radiculopathy will participate in this study. The patients will randomly be divided into two equal groups; the control group which received the selected exercise program and the study group received the same exercise training program in addition to High Tone Power Therapy, three times per week for four weeks. The evaluation methods are cervical joint position error test, neck disability index, Cervical range of motion (CROM) and visual analogue scale

ELIGIBILITY:
Inclusion Criteria:

* Their ages range from 35 to 50 years.
* Both sex
* With mild to moderate cervical disability according to the neck disability index
* Unilateral cervical radiculopathy for more than 6 months.
* Cervical radiculopathy due to disc prolapse (C5-C6) (C6-C7) mild to moderate or disc prolapse according to magnetic resonance image (MRI).
* Normal body mass index (18.5 - 24.99Kg/m2).

Exclusion Criteria:

* Any other musculoskeletal disorders of the spine or upper extremity
* Patients with any other Neurological deficits, psychiatric disease Cervical myelopathy, Cognitive problems, vertebral fractures and previous history of spine or cervical surgery.
* Neck pain with vertigo or with bilateral upper limbs referred pain.
* Clinical instability, recent trauma and vertebrobasilar insufficiency.
* Structural abnormalities of the spine, osteoporosis, and spasmodic torticollis.
* Inflammatory or other specific disorders of spina such as ankylosing spondylitis and rheumatoid arthritis

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
cervical joint position error test | four weeks
  The subject will be instructed to perform an active head rotation to one side, after which returns back to the neutral or starting head position.
  The test will be performed in a 3 trials in each direction
Neck disability index | four weeks
  includes 10 items as follows: Pain Intensity, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, and Recreation, with a score (0:5) for every point. The maximum score is 50, with the interpretation scoring (no disability = 0: 4, mild disability 5:14, moderate disability 15:24, severe disability 25: 34 and complete disability above 34
CROM | four weeks
  Cervical range of motion measured using CROM in different directions

SECONDARY OUTCOMES:
Visual analogue scale for pain (VAS-P) | four weeks
  is a method for measuring the intensity of pain on a horizontal straight line of fixed length (10 cm), as the left end of the line showed the greatest pain score & the right end showed the least pain scores, then the patient was asked to put a mark, on the line according to his/her pain sensation, with a higher score representing the higher level of pain

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 university, Giza, Giza Governorate, Egypt